CLINICAL TRIAL: NCT04637035
Title: Feasibility of Delivering a Supportive Oncology Care at Home Intervention for Hospitalized Patients With Cancer
Brief Title: Supportive Oncology Care at Home Post-Discharge
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Medically Home Group, Inc. (Unknown)
Responsible Party: Principal Investigator, Ryan Nipp, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-414
Record Dates: First submitted 2020-10-29; First posted 2020-11-19 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cancer
Keywords: Cancer; Home Care; Remote Monitoring
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Oncology Care at Home (Experimental): Participants will receive the Supportive Oncology Care at Home program for 14 days following their discharge from the hospital.
  The Supportive Oncology Care at Home intervention consists of three key components:
  * Daily monitoring of patient-reported symptoms, vital signs, and body weight.
  * Medically Home care based on algorithmic changes in patients' daily symptoms, vital signs, and body weight.
  * Structured communication with the oncology team regarding care delivered to ensure continuity of care.
  Interventions: Other: Supportive Oncology Care at Home

INTERVENTIONS:
Other: Supportive Oncology Care at Home — Intervention entailing remote monitoring of patients' symptoms, vital signs, and body weight with home-based care.

SUMMARY:
This study is evaluating if a program that involves remote monitoring and home-based care may improve the post-discharge care of recently hospitalized patients with advanced cancer.

The Supportive Oncology Care at Home intervention consists of three key components:

1. Remote patient monitoring (e.g. patient-reported symptoms, home-monitored vital signs and body weight);
2. A Medically Home care model for symptom assessment, evaluation, and management (e.g. triggers for phone calls and visits to patients' homes to address and manage any concerning issues identified);
3. Structured communication with the oncology team to ensure continuity of care.

DETAILED DESCRIPTION:
This is a single-arm pilot study of recently hospitalized patients with advanced cancer to assess the the feasibility of delivering a remote monitoring and home-based program, Supportive Oncology Care at Home, the acceptability and satisfaction with the Supportive Oncology Care at Home program, and changes in the quality of life and symptoms of patients who receive the Supportive Oncology Care at Home program.

Oncologists at the MGH Cancer Center developed the Supportive Oncology Care program to address the symptoms and frequent hospital visits that patients face as a result of their cancer and the treatment they receive.

The research study procedures include:

* Remote monitoring of symptoms, vital signs, and body weight
* Questionnaires asking about demographic information (e.g. gender, ethnicity, income) and participant experience with cancer (e.g. your quality of life, your symptoms)
* Interviews to assess participant impressions of the program
* Caregiver Interviews, Questionnaires and Surveys to assess caregiver impressions of the program and caregiver perceptions of participant symptoms while in the program
* Clinician Interviews and Questionnaires to assess impressions of the program
* Data collection from participant medical record.

Patients will take part in the program for two weeks following hospital discharge.

It is expected that between 75 and 110 people will enroll, including up to 30 patients, up to 30 caregivers, and up to 15 clinicians.

Medically Home Group, Inc. is supporting this research study by providing funding for this research study.

ELIGIBILITY:
Inclusion Criteria:

Patient Eligibility

* Age 18 or older
* Diagnosed with advanced cancer (defined as receiving treatment with palliative intent per chemotherapy order entry treatment intent designation and/or trial consent forms OR based on documentation in the oncology clinic notes for those not receiving chemotherapy)
* Admitted with an unplanned or non-elective hospitalization at Massachusetts General Hospital (MGH)
* Not requiring ICU-level care during their hospitalization
* Receiving care at the MGH Cancer Center
* Ability to read and respond to question in English
* Residing within 50 miles of MGH.

Caregiver Eligibility

* Relative or friend of eligible patient
* Verbally fluent in English
* Age 18 or older

Clinician Eligibility

-- Outpatient oncology physicians and advanced practice clinicians who care for patients that receive the Supportive Oncology Care at Home intervention

Exclusion Criteria:

Patient Exclusion

* Are admitted to the intensive care unit
* Have a high oxygen requirement (FIO2 > 0.40)
* Experience active angina or cardiac arrythmias
* Have a planned inpatient surgical or interventional procedure
* Have uncontrolled psychiatric illness or impaired cognition interfering with their ability to understand study procedures and provide written informed consent
* Are deemed ineligible for home-based care based on the inpatient oncology clinician assessment
* Are planning to be discharged to hospice or to any location other than their home

Caregiver Exclusion -- Caregivers who are unwilling or unable to participate in the study.

Clinician Exclusion

-- Clinicians who are unwilling or unable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of study enrollment | 2 years
  Proportion of patients who agree to participate in the study and sign informed consent.
Rates of completion of daily symptom assessment | 2 years
  Proportion of daily patient-reported symptom assessments completed throughout the study period.

SECONDARY OUTCOMES:
Rates of completion of daily vital signs | 2 years
  Proportion of daily vital signs completed throughout the study period.
Rates of completion of daily body weight | 2 years
  Proportion of daily reporting body weights completed throughout the study period.
Number of home visits required | Baseline to 2 weeks post-enrollment
  Number of home visits required, their average duration, the issues addressed at home, and the interventions delivered to patients at their home.
Duration of home visits | Baseline to 2 weeks post-enrollment
  Average duration of home visits required during the study period.
Issues addressed during home visits | Baseline to 2 weeks post-enrollment
  Issues addressed during home visit throughout the study period.
Interventions delivered during home visits | Baseline to 2 weeks post-enrollment
  Interventions delivered to patients at their home throughout the study period.
Number of phone calls required | Baseline to 2 weeks post-enrollment
  Number of phone calls required per patient.
Duration of phone calls | Baseline to 2 weeks post-enrollment
  Average duration of phone calls required for patients.
Number of emails required | Baseline to 2 weeks post-enrollment
  Number of emails from Medically Home to the primary oncology team.
Patient acceptability | 1 year
  Qualitative interview acceptability ratings from patients regarding usefulness, effectiveness, and relevance of the study.
Family caregiver acceptability | 1 year
  Qualitative interview acceptability ratings from caregivers regarding usefulness, effectiveness, and relevance of the study.
Clinician acceptability | 1 year
  Qualitative interview acceptability ratings from clinicians regarding usefulness, effectiveness, and relevance of the study.
Change in symptoms burden longitudinally throughout the study | Baseline to 2 weeks post-enrollment
  Change in symptom burden (assessed using Edmonton Symptom Assessment System-revised [ESAS-r], range 0-10 for each symptom with higher score indicating worse symptom burden) throughout the study.
Change in psychological distress score longitudinally throughout the study | Baseline to 2 weeks post-enrollment
  Change in psychological distress (assessed using Hospital Anxiety and Depression Scale [HADS], range 0-21 for scores of anxiety and depression with higher score indicating worse anxiety or depression) throughout the study.
Change in quality of life score longitudinally throughout the study | Baseline to 2 weeks post-enrollment
  Change in quality of life (assessed using Functional Assessment of Cancer Therapy-General [FACT-G] questionnaire, assessing physical, functional, emotional, and social well-being during the prior seven days, with total score ranging from 0-108 with higher scores indicating better quality of life) throughout the study.
Change in care satisfaction score longitudinally throughout the study | Baseline to 2 weeks post-enrollment
  Change in patient care satisfaction (assessed using the 16-item FAMCARE questionnaire [FAMCARE-P], range of 16-80 with higher score indicating higher care satisfaction) throughout the study.
Number of emergency department visits | Baseline up to one month post-enrollment
  The number of emergency department [ED] visits per patient.
Rates of emergency department visits | 1 year
  Proportion of patients needing an emergency department [ED] visit.
Number of urgent visits | Baseline up to one month post-enrollment
  The number of urgent visits to clinic per patient.
Rates of urgent visits | 1 year
  Proportion of patients needing an urgent visit to clinic.
Number of hospital readmissions | Baseline up to one month post-enrollment
  The number of hospital readmissions per patient.
Rates of hospital readmissions | 1 year
  Proportion of patients needing hospital readmission.
Length of hospital readmissions | Baseline up to one month post-enrollment
  The length of stay (LOS) per each hospital readmission for patients who are readmitted.
Days outside of hospital | Baseline to 2 weeks post-enrollment
  The proportion of days patients spent outside the hospital during the study period.
Hospitalization length of stay | Baseline to 2 weeks post-enrollment
  The index hospitalization length of stay (LOS).
Change in caregivers reports of patients' symptom burden longitudinally throughout the study | Baseline to 2 weeks post-enrollment
  Change in symptom burden (assessed using Edmonton Symptom Assessment System-revised [ESAS-r], range 0-10 for each symptom with higher score indicating worse symptom burden) throughout the study.
Concordance between caregiver and patient reports of patient symptom burden | Baseline to 2 weeks post-enrollment
  Difference in symptom burden (assessed using Edmonton Symptom Assessment System-revised [ESAS-r], range 0-10 for each symptom with higher score indicating worse symptom burden) between patients and caregivers throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan D Nipp, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Description: The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Nipp RD, Shulman E, Smith M, Brown PMC, Johnson PC, Gaufberg E, Vyas C, Qian CL, Neckermann I, Hornstein SB, Reynolds MJ, Greer J, Temel JS, El-Jawahri A. Supportive oncology care at home interventions: protocols for clinical trials to shift the paradigm of care for patients with cancer. BMC Cancer. 2022 Apr 9;22(1):383. doi: 10.1186/s12885-022-09461-z. PMID 35397575